CLINICAL TRIAL: NCT01338350
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled AZD5423 After Administration of Single and Multiple Ascending Doses in Healthy Male Japanese Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics After Single and Multiple Dosing of AZD5423 in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2340C00003
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; pharmacodynamics; AZD5423; Japanese
MeSH Terms: interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD5423
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5423 — Inhalation, suspension
  Arms: 1
Drug: Placebo — Inhalation, solution
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics and pharmacodynamic effects (24-hours plasma cortisol area under curve, plasma cortisol pre and post ACTH stimulation, dehydroepiandrosterone sulphate (DHEAS), osteocalcin and 24 hours urine cortisol) of AZD5423 following administration of single and multiple ascending doses in healthy male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male Japanese subjects aged 20 to 45 years with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms, from the day of dosing until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 18 and 27 kg/m2 and weight at least 50 kg and no more than 80 kg
* Be able to inhale from the I-nebⓇ according to given instruction

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of investigational product
* Any clinically significant abnormalities in clinical chemistry, haematology, urinalysis or physical examination results as judged by the investigators
* Any positive results on screening for serum hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV) and Syphilis

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability (AE, blood pressure, pulse, ECG, Body temp, Haematology, Clin Chemistry, Urinalysis, phys exam, lung function) of AZD5423 following administration of single and multiple ascending doses. | 10-14 days after last dose

SECONDARY OUTCOMES:
To characterise the single and multiple dose pharmacokinetics of AZD5423, and assess the dose proportionality, the time required to reach steady state and the degree of accumulation. | 72 hours after last dose
To investigate the pharmacodynamic effects (24-hours plasma cortisol AUC, plasma cortisol pre and post ACTH stimulation, DHEAS, osteocalcin and 24 hours urine cortisol) of AZD5423 following administration of single and multiple ascending doses. | 10-14 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Fukuoka, Japan

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1256&filename=D2340C00003.pdf